CLINICAL TRIAL: NCT00344097
Title: The Effects of Soy Protein Supplementation on Post-thoracotomy Pain
Brief Title: The Effects of Soy Protein on Post-thoracotomy Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21 AT003613
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Thoracotomy; Pain
Keywords: soy protein; pain; thoracotomy
MeSH Terms: conditions — Pain | interventions — Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Soy protein

SUMMARY:
This study seeks to determine whether soy protein supplements reduce the pain that often occurs following surgery for a lung tumor. Patients are randomized to receive either soy protein or milk protein prior to and following a thoracotomy for a lung tumor. We are especially interested in pain severity and pain medication use following surgery and will measure function and quality of life.

DETAILED DESCRIPTION:
Preclinical studies indicate that soy-containing diets suppress the development of pain behaviors and hyperalgesia seen following nerve injury and recent data indicate a similar protective effect of a diet high in soy protein in inflammatory and bone cancer pain models. These studies further indicate that soy exposure is only protective when administered in the period immediately preceding injury. Very few studies have directly studied the effects of soy-containing diets on pain sensitivity in humans, but one recent randomized clinical trial suggests that dietary soy supplementation may reduce pain due to osteoarthritis. The proposed study will examine whether a soy protein supplement reduces the pain commonly experienced following thoracotomy for lung surgery. This is a useful clinical model for studying the effects of soy protein supplementation on pain because the pain associated with surgery is quite severe and is one of the greatest concerns patients have about undergoing surgery. The growing recognition that greater acute pain leads to persistent pain following tissue healing underscores the importance of identifying viable strategies, including both non-pharmacological as well as pharmacological, for reducing the acute pain associated with surgery. Using a 2 group (soy protein supplementation vs. matched milk placebo supplementation) design, patients undergoing elective major open thoracotomy for segmentectomy, lobectomy, or bilobectomy will be randomly assigned to one of these two treatment groups. Patients will begin taking the soy/placebo supplement 2-3 days prior to thoracotomy and continue daily consumption of the supplement for an additional period following surgery. The feasibility/pilot study will examine the effects of soy supplementation on outcome measures during three post-operative time periods: 1) the immediate post-operative period; 2) during 2-12 weeks following surgery; and 3) during 14-24 weeks following surgery. Pain is the primary outcome domain of interest in this pilot study and measures will include pain severity ratings and pain medication use. Function and quality of life are the secondary outcome domains of interest and measures will include pain-related interference with daily activities, sleep, and health-related quality of life. Outcome measures will be collected bi-weekly throughout the study. The study aims to determine the feasibility and acceptability of soy supplementation in the period surrounding thoracotomy, determine level of adherence to soy supplementation over the 6-month period of follow-up, and estimate the effect size of soy supplementation relative to placebo in reducing significant pain following thoracotomy. The proposed study will provide the necessary groundwork to move towards such a larger randomized trial to evaluate the pain-reducing effects of soy protein supplementation following thoracotomy.

ELIGIBILITY:
Inclusion criteria: 1) undergoing major elective thoracotomy through a classic incision, including segmentectomy, lobectomy, or wedge resection, 2) for women, a negative mammogram within the past year; 3) for women using oral contraceptives or hormone replacement therapy, the agreement to hold steady dosing of these medications for the duration of the study; and 4) ability to comprehend the consent information and to complete all study assessments.

Exclusion criteria: 1) age less than 18 years, 2) current alcohol or substance abuse/dependence; 3) delirium, dementia, or cognitive impairment (MMSE < 24; (23)); 4) use of analgesics (other than aspirin or non-steroidal anti-inflammatories) for a condition other than the reason for surgery; 5) milk or soy allergy; 6) lactose intolerance; 7) pre-operative chest pain; 8) women with a history of breast cancer; or 9) [use of an antibiotic within 3 months prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
pain severity
pain medication use

SECONDARY OUTCOMES:
function
health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Haythornthwaite, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States